CLINICAL TRIAL: NCT05686850
Title: Non-Invasive Ventilation Versus High-flow Nasal Oxygen for Post-extubation Respiratory Failure in Intensive Care Units: a Multicenter, Randomized, Controlled Trial
Brief Title: Non-Invasive Ventilation Versus High-flow Nasal Oxygen in Intensive Care Units
Acronym: VENTILO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VENTILO Trial; 2022-A02189-34 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Post Extubation Respiratory Failure
Keywords: Respiratory Failure; post-Extubation; Intubation; Non-invasive ventilation; High-Flow nasal oxygen
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Flow Oxygen (Active Comparator): Patients assigned to the control group will be continuously treated by high-flow nasal oxygen during the 48 hours following randomization
  Interventions: Procedure: High-Flow Oxygen
- NIV alternating with High-Flow Oxygen (Experimental): Patients assigned to the intervention group will be treated with curative NIV alternating with high-flow nasal oxygen during the 48 hours following randomization
  Interventions: Procedure: High-Flow Oxygen; Procedure: Non invasive ventilation

INTERVENTIONS:
Procedure: High-Flow Oxygen — Humidified and heated oxygen with a gas flow at least 50 L/min through nasal cannula
Procedure: Non invasive ventilation — NIV will be carried out in pressure-support mode with a minimal pressure-support level of 5 cmH2O targeting a tidal volume around 6 to 8 mL/kg of predicted bodyweight, a positive end-expiratory pressure (PEEP) level at least 8 cm H2O, and FiO2 adjusted to obtain adequate oxygenation
  Arms: NIV alternating with High-Flow Oxygen

SUMMARY:
In intensive care units (ICUs), around 20% of patients experience respiratory failure after planned extubation. Nearly 40-50% of them eventually require reintubation with subsequently high mortality rates reaching 30-40%. NIV used as rescue therapy to treat post-extubation respiratory failure could increase the risk of death. However, NIV may avoid reintubation in a number of cases, and recent large-scale clinical trials on extubation have shown that around 40 to 50% of patients with post-extubation respiratory failure are actually treated with NIV. Whereas high-flow nasal oxygen has never been specifically studied for management of post-extubation respiratory failure, this respiratory support could also in this setting constitute an alternative to standard oxygen or NIV. Given the best noninvasive respiratory support strategy in patients with post-extubation respiratory failure remains unknown, we have decided to assess whether NIV alternating with high-flow nasal oxygen as compared to high-flow nasal oxygen alone may decrease mortality of patients in ICUs with post-extubation respiratory failure.

DETAILED DESCRIPTION:
In intensive care units (ICUs), around 20% of patients experience respiratory failure after planned extubation (defined as removal of endotracheal tube after weaning from the ventilator). Nearly 40-50% of them eventually require reintubation with subsequently high mortality rates reaching 30-40%.Consequently, a noninvasive respiratory support strategy aiming at avoiding reintubation deserves consideration. Whereas prophylactic use of non-invasive ventilation (NIV) applied immediately after extubation may prevent respiratory failure, NIV used as rescue therapy to treat established post-extubation respiratory failure could increase the risk of death. The largest clinical trial conducted to date by Esteban and colleagues showed greater mortality with NIV than with standard oxygen. The only factor explaining the deleterious effects of NIV was that the time before reintubation was markedly longer than with standard oxygen, suggesting that NIV may worsen the outcome by delaying reintubation. No further large-scale clinical trial has been performed after this study and thereby, the most recent international clinical practice guidelines suggest that NIV should not be used in this setting. However, recent large-scale clinical trials on extubation have shown that around 40 to 50% of patients with post-extubation respiratory failure are actually treated with NIV. Indeed, NIV as rescue therapy may avoid reintubation in a number of cases, especially in patients with underlying chronic lung disease. In a recent post-hoc analysis focusing on 146 patients with established post-extubation respiratory failure, we found that mortality was 18% with NIV and 29% with high flow nasal oxygen alone (difference, - 11% [95% CI, -25% to 2%]; p=0.12). Mortality rates were even significantly lower with NIV than with high-flow nasal oxygen alone in patients with hypercapnia, suggesting that after all, NIV might not increase the risk of death. To explain the discrepancies with the Esteban study, the time interval between NIV initiation and reintubation was markedly shorter in our study (5 hours in median vs. 12) and predefined criteria for reintubation were established in order to minimize the risk of delayed intubation. Moreover, all participating centers had extensive experience in NIV which was not the case in the previous trial. Whereas high-flow nasal oxygen has never been specifically studied for management of post-extubation respiratory failure, this respiratory support could in this setting constitute an alternative to standard oxygen or NIV. High-flow nasal oxygen is increasingly used after extubation in order to prevent post-extubation respiratory failure, and its beneficial effects have been reported in treatment of acute respiratory failure. To date, the best noninvasive respiratory support strategy in patients with post-extubation respiratory failure remains unknown. However, high-flow nasal oxygen could be included among reference respiratory supports whereas standard oxygen would be considered as a suboptimal strategy after extubation in ICUs.Thereby, we have decided to assess whether NIV alternating with high-flow nasal oxygen as compared to high-flow nasal oxygen alone may decrease mortality of patients in ICUs with post-extubation respiratory failure.

To do that, we propose to conduct a prospective multicenter randomized controlled open-label trial comparing these 2 strategies of noninvasive respiratory support in patients with post-extubation respiratory failure in ICUs. Patients included will be randomized as early as possible after the onset of respiratory failure and will be assigned to one of the 2 following groups, with a 1:1 ratio: high-flow nasal oxygen group treated by high-flow nasal oxygen alone, or NIV group treated by NIV alternating with high-flow nasal oxygen. As NIV may be more effective in hypercapnic patients, randomization will be stratified according to the PaCO2 level measured on blood gas performed at inclusion with the aim at ensuring a balanced allocation of hypercapnic patients (PaCO2 > 45 mmHg) among the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Duration of invasive mechanical ventilation of more than 24h in the ICU before extubation.
* Post-extubation respiratory failure occurring within the first 7 days after extubation (see criteria below). As in several previous studies, post-extubation respiratory failure will be defined by the presence of the 2 following criteria combining a clinical criterion and a blood gas criterion:

  * Clinical criterion persisting for at least 30 minutes: a respiratory rate exceeding 25 breaths per minute or clinical signs of respiratory distress with increased accessory muscle activity.
  * Blood gas criterion: Hypoxemia defined as PaO2/FiO2 ratio below 150 mm Hg or respiratory acidosis defined as pH below 7.35 units and PaCO2 above 45 mm Hg. For patients under standard oxygen, FiO2 will calculated according to the following formula: FiO2 = 0.21 + 0.03 x (oxygen flow L/min).
* Informed consent from the relatives or the patient himself, or emergency inclusion procedure in case of inability of patient or proxy to give consent.

Exclusion Criteria:

* NIV at home
* ICU admission for peripheral neuromuscular disease type Guillain-Barré syndrome or myasthenia gravis.
* Upper airway obstruction as main reason for post-extubation respiratory failure
* Urgent need for reintubation (respiratory or cardiac arrest, respiratory pauses with loss of consciousness or gasping for air, or severe hypoxemia defined as SpO2 lower than 90% despite maximal oxygen support)
* Altered consciousness (Glasgow coma scale < 12)
* Unplanned extubation (accidental or self-extubation)
* Do-not-reintubate order at time of respiratory failure
* Patient previously included in the study
* People under protection (minors, persons deprived of liberty by a judicial or administrative decision, adults under law protection)
* Patient not affiliated to health care system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2028-02-27 (Estimated); Study Completion 2028-08-27 (Estimated)

PRIMARY OUTCOMES:
Mortality at 28 days after post-extubation respiratory failure | Day 28
  Death between post-extubation respiratory failure and 28 days after post-extubation respiratory failure

SECONDARY OUTCOMES:
Time to death between randomization and day 28 | Day 28
  Death between randomization and day 28
Reintubation within the 48 hours, 7 days and 28 days following post-extubation respiratory failure | Hour 48 Day 7 and Day 28
  Reintubation rates within the 48 hours, 7 days and 28 days following respiratory failure
Ventilator-free days at day 28, | Day 28
  number of days alive and without invasive mechanical ventilation between randomization (day 1) and day 28.
Length of stay in ICU and length of stay in hospital. | Day 90
  Length of stay in ICU and length of stay in hospital in days
Mortality in ICU, in hospital and at day 90. | Day 90
  Number of death in ICU, in hospital and at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud W. THILLE, PhD, Principal Investigator — CHU Poitiers
Locations (1):
- CHU Poitiers, Poitiers, France